CLINICAL TRIAL: NCT03487159
Title: Using the Non Invasive Technology Magnetic Resonance Elastography for the Diagnosis of Liver Fibrosis Stage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Prof. Ziv Ben-Ari MD (Other Government)
Responsible Party: Sponsor-Investigator, Prof. Ziv Ben-Ari MD, Head of Liver Diseases Center, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEBA-17-4749-ZBA-CTIL
Record Dates: First submitted 2018-02-19; First posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Intervention Model Description: The study model includes 2 study arms:
  1. Patients with chronic liver diseases who will undergo a routine liver biopsy, Shear Wave elastography and the MRE in order to evaluate the liver fibrosis stage.
  2. Patients with chronic liver diseases who will undergo a routine Shear Wave elastography and the MRE in order to evaluate the liver fibrosis stage.
  Demographic and clinical information will be collected from the patient's medical files.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liver biopsy ,Elastography and MRE (Other): Performance of routine Liver biopsy,Shear Wave Elastography and investigational MRE (Magnetic Resonance Elastography) in order to evaluate liver fibrosis stage.
  Interventions: Device: MRE (Magnetic Resonance Elastography)
- Elastography and MRE (Other): Performance of routine Shear Wave Elastography and investigational MRE (Magnetic Resonance Elastography) in order to evaluate liver fibrosis stage.
  Interventions: Device: MRE (Magnetic Resonance Elastography)

INTERVENTIONS:
Device: MRE (Magnetic Resonance Elastography) — The device is using to evaluate liver fibrosis stage

SUMMARY:
This study evaluates the ability of Magnetic Resonance Elastography non invasive technology to identify the liver fibrosis stage in patients with chronic liver diseases compared to Shear Wave Elastography and/or Liver Biopsy.

DETAILED DESCRIPTION:
Recent advances in magnetic resonance imaging (MRI) of the liver have led to improvements in diagnosis of chronic liver diseases. Detection and staging of liver fibrosis has become important; however, until about the last decade, it depended on an invasive liver biopsy. Liver biopsy is limited by high cost, low patient acceptance, interobserver variability during microscopic evaluation, sampling error, poor reproducibility, and, importantly, an invasive nature with a complication rate of 3% and a mortality rate of 0.03%. With the emergence of elastography techniques, the need for liver biopsy has rapidly diminished for diagnosis of clinically significant liver fibrosis. Magnetic Resonance Elastography has gained increasing popularity in recent years, in large part due to its higher technical success and ability to overcome some of the weaknesses of ultrasound-based methods for assessing liver fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic liver diseases

Exclusion Criteria:

* Patients who don't have chronic liver diseases

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Liver Biopsy Result for liver fibrosis grade | Patient will undergo Liver biopsy once during 1 year of the study.
  Liver Fibrosis score measured by Metavir scale .The Metavir score grades the degree of fibrosis on a 5-point scale from 0 to 4. The activity, which is the amount of inflammation (specifically, the intensity of necro-inflammatory lesions), is graded on a 4-point scale from A0 to A3.
  Fibrosis score:
  F0 = no fibrosis F1 = portal fibrosis without septa F2 = portal fibrosis with few septa F3 = numerous septa without cirrhosis F4 = cirrhosis
  Activity score:
  A0 = no activity A1 = mild activity A2 = moderate activity A3 = severe activity Liver biopsy will be perfomed only according to physician recommendation.
Magnetic Resonance Elastography (MRE) Result for liver fibrosis grade | Patient will undergo Magnetic Resonance Elastography (MRE) once during 1 year of the study.
  Liver Fibrosis score determined by liver stiffness in 4 fibrosis grades: >1=any fibrosis, >2=significant fibrosis, >3=advanced fibrosis, 4=cirrhosis
Shear Wave Elastography Result for liver fibrosis grade | Patient will undergo Shear Wave Elastography once during 1 year of the study.
  Liver Fibrosis score determined by liver stiffness in in 5 fibrosis grades: 0=no fibrosis, >1=any fibrosis, >2=significant fibrosis, >3=advanced fibrosis, 4=cirrhosis

CONTACTS AND LOCATIONS:
Overall Officials: Ziv Ben-Ari, MD, Principal Investigator — Liver Diseases Center, Sheba M.C
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No